CLINICAL TRIAL: NCT02064439
Title: Reduced-dosed Rivaroxaban and Standard-dosed Rivaroxaban Versus ASA in the Long-term Prevention of Recurrent Symptomatic Venous Thromboembolism in Patients With Symptomatic Deep-vein Thrombosis and/or Pulmonary Embolism
Brief Title: Reduced-dosed Rivaroxaban in the Long-term Prevention of Recurrent Symptomatic VTE(Venous Thromboembolism)
Acronym: EinsteinChoice
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 16416; 2013-000619-26 (EudraCT Number)
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Pulmonary Embolism; Thromboembolism; Thrombosis; Venous Thrombosis; Venous Thromboembolism
Keywords: deep vein thrombosis; pulmonary embolism; long-term prevention of recurrent symptomatic VTE
MeSH Terms: conditions — Pulmonary Embolism; Thromboembolism; Thrombosis; Venous Thrombosis; Venous Thromboembolism | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Rivaroxaban 10 mg once daily for 12 months
  Interventions: Drug: BAY 59-7939
- Arm 2 (Experimental): Rivaroxaban 20 mg once daily for 12 months
  Interventions: Drug: BAY 59-7939
- Arm 3 (Active Comparator): ASA (Acetylsalicylic Acid) 100 mg once daily for 12 months
  Interventions: Drug: ASA

INTERVENTIONS:
Drug: BAY 59-7939 — 10 mg tablet once daily for 12 months
  Arms: Arm 1
Drug: BAY 59-7939 — 20 mg tablet once daily for 12 months
  Arms: Arm 2
Drug: ASA — 100 mg tablet once daily for 12 months
  Arms: Arm 3

SUMMARY:
This is a multicenter, randomized, double-blind, event-driven, superiority study for efficacy.

Patients with confirmed symptomatic DVT (Deep Vein Thrombosis) or PE (Pulmonary embolism) who completed 6 or 12 months of treatment of anticoagulation are eligible for this trial

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed symptomatic PE and/or DVT who have been treated for 6 to 12 months and did not interrupt anticoagulation for longer than 1 week

Exclusion Criteria:

* Legal lower age limitations (country specific) Indication for therapeutic-dosed anticoagulants Indication for antiplatelet therapy or a conventional non-steroid anti-inflammatory drug (NSAID) Hepatic disease which is associated with coagulopathy leading to a clinically relevant bleeding risk Calculated creatinine clearance < 30 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3365 (Actual)
Dates: Start 2014-03-05 (Actual); Primary Completion 2016-09-22 (Actual); Study Completion 2016-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (224):
- United States (22):
  - Beverly Hills, California
  - La Jolla, California
  - Ventura, California
  - Denver, Colorado
  - Jacksonville, Florida
  - Columbus, Georgia
  - Joliet, Illinois
  - Rockport, Maine
  - Boston, Massachusetts
  - Detroit, Michigan
  - Butte, Montana
  - Las Vegas, Nevada
  - Raleigh, North Carolina
  - Columbus, Ohio
  - Toledo, Ohio
  - Philadelphia, Pennsylvania
  - San Antonio, Texas
  - Fredericksburg, Virginia
  - Bellevue, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Tacoma, Washington
- Australia (12):
  - Garran, Australian Capital Territory
  - Concord, New South Wales
  - Kogarah, New South Wales
  - Lismore, New South Wales
  - Randwick, New South Wales
  - St Leonards, New South Wales
  - Westmead, New South Wales
  - Brisbane, Queensland
  - Clayton, Victoria
  - Box Hill
  - Melbourne
  - Redcliffe
- Austria (3):
  - Graz, Styria
  - Innsbruck, Tyrol
  - Vienna
- Belgium (4):
  - Aalst
  - Bruxelles - Brussel
  - Hasselt
  - Leuven
- Brazil (7):
  - Belo Horizonte, Minas Gerais
  - Porto Alegre, Rio Grande do Sul
  - Campinas, São Paulo
  - Santo André, São Paulo
  - São Paulo, São Paulo
  - Rio de Janeiro
  - São Paulo
- Canada (9):
  - Edmonton, Alberta
  - Victoria, British Columbia
  - Saint John, New Brunswick
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Montreal, Quebec
  - Saint-Jérôme, Quebec
- China (24):
  - Fuzhou, Fujian
  - Guangzhou, Guangdong
  - Nanning, Guangxi
  - Shijiazhuang, Hebei
  - Harbin, Heilongjiang
  - Wuhan, Hubei
  - Changsha, Hunan
  - Nantong, Jiangsu
  - Suzhou, Jiangsu
  - Changchun, Jilin
  - Shengyang, Liaoning
  - Shenyang, Liaoning
  - Yinchuan, Ningxia
  - Xi'an, Shaanxi
  - Jinan, Shandong
  - Qingdao, Shandong
  - Taiyuan, Shanxi
  - Chengdu, Sichuan
  - Kunming, Yunnan
  - Hangzhou, Zhejiang
  - Wenzhou, Zhejiang
  - Beijing
  - Shanghai
  - Tianjin
- Czechia (6):
  - Kladno
  - Liberec
  - Litomyšl
  - Ostrava
  - Prague
  - Ústí nad Labem
- Denmark (7):
  - Aarhus N
  - Copenhagen
  - Glostrup Municipality
  - Hellerup
  - Herning
  - København NV
  - Svendborg
- France (21):
  - Angers
  - Arras
  - Besançon
  - Bois-Guillaume
  - Brest
  - Castelnau-le-Lez
  - Clermont-Ferrand
  - Colombes
  - Dijon
  - Grenoble
  - Le Kremlin-Bicêtre
  - Le Mans
  - Limoges
  - Nice
  - Paris
  - Quimper
  - Saint-Etienne
  - Strasbourg
  - Toulon
  - Toulouse
  - Vernon
- Germany (10):
  - Heidelberg, Baden-Wurttemberg
  - München, Bavaria
  - Darmstadt, Hesse
  - Witten, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Dresden, Saxony
  - Magdeburg, Saxony-Anhalt
  - Erfurt, Thuringia
  - Berlin
  - Karlsbad
- Hungary (10):
  - Baja
  - Budapest
  - Debrecen
  - Gyula
  - Kecskemét
  - Miskolc
  - Pécs
  - Szentes
  - Szombathely
  - Zalaegerszeg
- Israel (8):
  - Afula
  - Haifa
  - Holon
  - Kfar Saba
  - Nahariya
  - Petah Tikva
  - Safed
  - Tel Aviv
- Italy (8):
  - Chieti, Abruzzo
  - Cosenza, Calabria
  - Piacenza, Emilia-Romagna
  - Reggio Emilia, Emilia-Romagna
  - Varese, Lombardy
  - Perugia, Umbria
  - Padua, Veneto
  - Treviso, Veneto
- Mexico (7):
  - León, Guanajuato
  - Guadalajara, Jalisco
  - Monterrey, Nuevo León
  - Xalapa, Veracruz
  - Mérida, Yucatán
  - Aguascalientes
  - Chihuahua City
- Netherlands (10):
  - Alkmaar
  - Almere Stad
  - Amsterdam
  - Assen
  - Dordrecht
  - Groningen
  - Hoofddorp
  - Maastricht
  - Sittard
  - Zwolle
- New Zealand (4):
  - Auckland
  - Christchurch
  - Palmerston North
  - Wellington
- Norway (2):
  - Fredrikstad
  - Oslo
- Quezon City, Philippines
- Poland (5):
  - Bialystok
  - Bydgoszcz
  - Poznan
  - Warsaw
  - Wroclaw
- Russia (8):
  - Barnaul
  - Moscow
  - Novosibirsk
  - Rostov-on-Don
  - Ryazan
  - Saint Petersburg
  - Sochi
  - Tver'
- South Africa (6):
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Pretoria West, Gauteng
  - Roodepoort, Gauteng
  - Worcester, Western Cape
  - Bloemfontein
- South Korea (4):
  - Donggu, Gwangju Gwang''yeogsi
  - Busan
  - Daegu
  - Seoul
- Spain (5):
  - Torrevieja, Alicante
  - L'Hospitalet de Llobregat, Barcelona
  - San Sebastián de los Reyes, Madrid
  - Girona
  - Madrid
- Sweden (2):
  - Gothenburg
  - Kristianstad
- Switzerland (6):
  - Basel, Canton of Basel-City
  - Lausanne, Canton of Vaud
  - Bern
  - Fribourg
  - Geneva
  - Lucerne
- Taiwan (3):
  - New Taipei City
  - Taichung
  - Taipei
- Thailand (2):
  - Bangkok
  - Khon Kaen
- Istanbul, Turkey (Türkiye)
- United Kingdom (5):
  - Plymouth, Devon
  - Hull, Humberside
  - Newcastle upon Tyne, Tyne and Wear
  - Cardiff
  - London
- Vietnam (2):
  - Hà Nội
  - Ho Chi Minh City

REFERENCES:
- [Background] Weitz JI, Bauersachs R, Beyer-Westendorf J, Bounameaux H, Brighton TA, Cohen AT, Davidson BL, Holberg G, Kakkar A, Lensing AW, Prins M, Haskell L, van Bellen B, Verhamme P, Wells PS, Prandoni P; EINSTEIN CHOICE Investigators. Two doses of rivaroxaban versus aspirin for prevention of recurrent venous thromboembolism. Rationale for and design of the EINSTEIN CHOICE study. Thromb Haemost. 2015 Aug 31;114(3):645-50. doi: 10.1160/TH15-02-0131. Epub 2015 May 21. PMID 25994838
- [Derived] Dobesh PP, Volkl AA, Pap AF, Damaraju CV, Levitan B, Yuan Z, Amin AN. Benefit-Risk Assessment of Rivaroxaban in Older Patients With Nonvalvular Atrial Fibrillation or Venous Thromboembolism. Drugs Aging. 2025 May;42(5):469-484. doi: 10.1007/s40266-025-01192-7. Epub 2025 Mar 31. PMID 40163217
- [Derived] Yamada N, Fu W, Shi Z, Park KH, Kim HS, Dai X, Lensing AW, Pap AF, Kohno T, Tajima T, Watakabe T, Mitsumori T. Risk of recurrent venous thromboembolism and major bleeding according to risk factor profiles in Asian patients: a subgroup analysis EINSTEIN-Extension and EINSTEIN-CHOICE. Thromb J. 2024 Jun 6;22(1):48. doi: 10.1186/s12959-024-00609-4. PMID 38844941
- [Derived] Flumignan CD, Nakano LC, Baptista-Silva JC, Flumignan RL. Antiplatelet agents for the treatment of deep venous thrombosis. Cochrane Database Syst Rev. 2022 Jul 25;7(7):CD012369. doi: 10.1002/14651858.CD012369.pub2. PMID 35876829
- [Derived] Weitz JI, Lensing AWA, Prins MH, Bauersachs R, Beyer-Westendorf J, Bounameaux H, Brighton TA, Cohen AT, Davidson BL, Decousus H, Freitas MCS, Holberg G, Kakkar AK, Haskell L, van Bellen B, Pap AF, Berkowitz SD, Verhamme P, Wells PS, Prandoni P; EINSTEIN CHOICE Investigators. Rivaroxaban or Aspirin for Extended Treatment of Venous Thromboembolism. N Engl J Med. 2017 Mar 30;376(13):1211-1222. doi: 10.1056/NEJMoa1700518. Epub 2017 Mar 18. PMID 28316279

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total 3439 participants were screened at 244 sites in 31 countries from 05-Mar-2014 (First Patient First Visit) to 15-Mar-2016 (Last Patient First Visit).
Pre-assignment Details: Of the 3439 participants screened 43 did not complete screening. Thus, 3396 participants were randomly assigned to treatment, 31 of the randomized participants never received study medication because either withdrew consent or were withdrawn from the study based on protocol violations.
Groups:
- Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD: Participants were randomized, stratified by country and by index event, to receive rivaroxaban 10 mg tablet or matching placebo once daily (OD) with food for 12, or 9 to less than 12, or 6 months depending on the date of randomization. Treatment of all participants stopped 6 months after the last participant was randomized.
- Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD: Participants were randomized, stratified by country and by index event, to receive rivaroxaban 20 mg tablet or matching placebo OD with food for 12, or 9 to less than 12, or 6 months depending on the date of randomization. Treatment of all participants stopped 6 months after the last participant was randomized.
- Acetylsalicylic (ASA) 100 mg, OD: Participants were randomized, stratified by country and by index event, to receive ASA 100 mg tablet or matching placebo OD with food for 12, or 9 to less than 12, or 6 months depending on the date of randomization. Treatment of all participants stopped 6 months after the last participant was randomized.
Period: Overall Study
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD | Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD | Acetylsalicylic (ASA) 100 mg, OD
Started | 1127 (Full Analysis Set (FAS), randomized and received study medication) | 1107 (FAS, randomized and received study medication) | 1131 (FAS, randomized and received study medication)
Completed | 984 | 969 | 949
Not Completed | 143 | 138 | 182
Not completed — Adverse Event | 51 | 47 | 46
Not completed — Death | 0 | 2 | 3
Not completed — Withdrawal by Subject | 29 | 18 | 26
Not completed — Protocol Violation | 3 | 5 | 3
Not completed — Lost to Follow-up | 1 | 3 | 4
Not completed — Non-compliance with study medication | 21 | 19 | 23
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Logistical difficulties | 6 | 5 | 2
Not completed — Efficacy outcome reached | 18 | 16 | 57
Not completed — Safety outcome reached | 12 | 20 | 10
Not completed — Other | 2 | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD | Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD | Acetylsalicylic (ASA) 100 mg, OD | Total
Number analyzed (Participants) | 1127 | 1107 | 1131 | 3365
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (14.7) | 57.9 (14.7) | 58.8 (14.7) | 58.5 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 507 | 505 | 488 | 1500
  Male | 620 | 602 | 643 | 1865
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 31 | 30 | 92
  Not Hispanic or Latino | 892 | 899 | 889 | 2680
  Unknown or Not Reported | 204 | 177 | 212 | 593
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2 | 4
  Asian | 161 | 159 | 159 | 479
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2 | 4
  Black or African American | 41 | 49 | 36 | 126
  White | 786 | 772 | 786 | 2344
  More than one race | 1 | 0 | 5 | 6
  Unknown or Not Reported | 135 | 126 | 141 | 402

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With the Composite of Fatal or Non-fatal Symptomatic Recurrent Venous Thromboembolism
Description: The primary efficacy outcomes (i.e., recurrent venous thromboembolism [VTE] defined as composite of fatal or non-fatal symptomatic recurrent VTE, including unexplained death for which pulmonary embolism [PE] could not be ruled out) as confirmed by the central independent adjudication committee (CIAC) were considered up to the end of the individual intended duration of treatment.
  Incidence of the composite of the primary and secondary efficacy outcome and its components are based on the first occurrence to participant.
Time Frame: Up to 12 months, at least 6 months
Measure: Number; unit: participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD | Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD | Acetylsalicylic (ASA) 100 mg, OD
Number analyzed (Participants) | 1127 | 1107 | 1131
participants
  Composite | 13 | 17 | 50
  Symptomatic recurrent Deep vein thrombosis (DVT) | 8 | 9 | 29
  Symptomatic recurrent PE | 5 | 6 | 19
  Death (PE) | 0 | 0 | 1
  Death (unexplained and PE cannot be ruled out) | 0 | 2 | 1
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD vs Acetylsalicylic (ASA) 100 mg, OD; Statistical analysis was performed on the first occurrence of the composite outcome; Test type: Superiority or Other; p = 0.0001, Wald test — P-value and hazard ratio estimates based on stratified proportional hazards model, with stratification based index event (DVT or PE with or without DVT); Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.20 to 0.59]
Statistical Analysis 2: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD vs Acetylsalicylic (ASA) 100 mg, OD; Statistical analysis was performed on the first occurrence of the composite outcome; Test type: Superiority or Other; p < 0.0001, Wald test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.26, 98% CI 2-sided [0.14 to 0.47]
Statistical Analysis 3: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD vs Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD; Statistical analysis was performed on the first occurrence of the composite outcome; Test type: Superiority or Other; p = 0.4328, Wald test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [0.65 to 2.75]

2. Primary Outcome: Number of Participants With First Treatment-emergent Major Bleeding
Description: The principal safety outcome was major bleeding which was defined according to the criteria of the International Society on Thrombosis and Hemostasis (ISTH) as clinically overt bleeding and associated with a fall in hemoglobin of 2 gram per deciliter (g/dL) or more, or leading to a transfusion of 2 or more units of packed red blood cells or whole blood, or occurring in a critical site, e.g. intracranial, intraspinal, intraocular, pericardial, intra articular, intramuscular with compartment syndrome, retroperitoneal, or contributing to death.
  Incidence of the composite of the primary and secondary efficacy outcome and its components are based on the first occurrence to participant.
Time Frame: Up to 12 months, at least 6 months
Measure: Number; unit: participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD | Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD | Acetylsalicylic (ASA) 100 mg, OD
Number analyzed (Participants) | 1127 | 1107 | 1131
participants
  Any major bleeding | 5 | 6 | 3
  Fatal bleeding | 0 | 1 | 1
  Non-fatal critical organ bleed | 2 | 4 | 1
  Non-fatal non-critical organ bleeding | 3 | 1 | 1
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD vs Acetylsalicylic (ASA) 100 mg, OD; Statistical analysis was performed on the first occurrence of the composite outcome; Test type: Superiority or Other; p = 0.3235, Wald test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 2.01, 95% CI 2-sided [0.50 to 8.04]
Statistical Analysis 2: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD vs Acetylsalicylic (ASA) 100 mg, OD; Statistical analysis was performed on the first occurrence of the composite outcome; Test type: Superiority or Other; p = 0.5005, Wald test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [0.39 to 6.84]
Statistical Analysis 3: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD vs Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD; Statistical analysis was performed on the first occurrence of the composite outcome; Test type: Superiority or Other; p = 0.7337, Wald test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.37 to 4.03]

3. Secondary Outcome: Number of Participants With the Composite of the Primary Efficacy Outcome, Myocardial Infarction, Ischemic Stroke or Systemic Non-CNS Embolism
Description: The secondary efficacy outcome is the composite of the primary efficacy outcome, myocardial infarction (MI), ischemic stroke or non-central nervous system (CNS) systemic embolism. Incidence of the composite of the primary and secondary efficacy outcome and its components are based on the first occurrence to participant.
Time Frame: Up to 12 months, at least 6 months
Measure: Number; unit: participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD | Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD | Acetylsalicylic (ASA) 100 mg, OD
Number analyzed (Participants) | 1127 | 1107 | 1131
participants
  Composite | 18 | 19 | 56
  Ischemic stroke | 4 | 2 | 2
  Non-CNS systemic embolism | 1 | 0 | 1
  Myocardial infarction | 0 | 1 | 4
  Symptomatic recurrent DVT | 8 | 9 | 29
  Symptomatic recurrent PE | 5 | 6 | 18
  Death (PE) | 0 | 0 | 1
  Death (unexplained and PE cannot be ruled out) | 0 | 1 | 1
  Death (cardiovascular: myocardial infarction) | 0 | 0 | 0
  Death (cardiovascular: ischemic stroke) | 0 | 0 | 0
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD vs Acetylsalicylic (ASA) 100 mg, OD; Statistical analysis was performed on the first occurrence of the composite outcome; Test type: Superiority or Other; p < 0.0001, Wald test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.20 to 0.57]
Statistical Analysis 2: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD vs Acetylsalicylic (ASA) 100 mg, OD; Statistical analysis was performed on the first occurrence of the composite outcome; Test type: Superiority or Other; p < 0.0001, Wald test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.32, 95% CI 2-sided [0.19 to 0.54]
Statistical Analysis 3: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD vs Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD; Statistical analysis was performed on the first occurrence of the composite outcome; Test type: Superiority or Other; p = 0.8172, Wald test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.57 to 2.06]

4. Secondary Outcome: Number of Participants With Non-major Bleeding Associated With Study Drug Interruption for > 14 Days
Description: The secondary safety outcome was clinically relevant non-major (CRNM) bleeding, which was adjudicated by the CIAC using the ASA criteria: the bleeding was non-major and the bleeding was associated with a study medication interruption of more than 14 days.
Time Frame: Up to 12 months, at least 6 months
Measure: Number; unit: participants
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD | Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD | Acetylsalicylic (ASA) 100 mg, OD
Number analyzed (Participants) | 1127 | 1107 | 1131
participants | 12 | 17 | 12
Statistical Analysis 1: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD vs Acetylsalicylic (ASA) 100 mg, OD; Test type: Superiority or Other; p = 0.3318, Wald test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.44, 95% CI 2-sided [0.69 to 3.02]
Statistical Analysis 2: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD vs Acetylsalicylic (ASA) 100 mg, OD; Test type: Superiority or Other; p = 0.9726, Wald test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.44 to 2.20]
Statistical Analysis 3: Comparison: Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD vs Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD; Test type: Superiority or Other; p = 0.3137, Wald test — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.46, 95% CI 2-sided [0.70 to 3.06]

ADVERSE EVENTS:
Time Frame: From after start of study medication but not more than 2 days after stop of study medication.
Arm/Group | Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD | Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD | Acetylsalicylic (ASA) 100 mg, OD
Serious Adverse Events (participants affected / at risk) | 78/1127 | 82/1107 | 79/1131
Other Adverse Events (participants affected / at risk) | 40/1127 | 35/1107 | 38/1131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD (N=1127) | Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD (N=1107) | Acetylsalicylic (ASA) 100 mg, OD (N=1131)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis constrictive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Cushing's syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Corneal degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis relapsing (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertrophic anal papilla (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colon dysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0)
Overlap syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Plasmodium falciparum infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 5 (6) | 3 (3)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urethral abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (6) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 2 (3) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Borrelia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Stomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Cystoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
B-lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 5 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cervix carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oesophageal carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 1 (1)
Cervix warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Malignant glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Ovarian cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Axonal neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (2)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Meningioma surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rivaroxaban (Xarelto, BAY59-7939) 10 mg, OD (N=1127) | Rivaroxaban (Xarelto, BAY59-7939) 20 mg, OD (N=1107) | Acetylsalicylic (ASA) 100 mg, OD (N=1131)
Atrial fibrillation (Cardiac disorders) | 6 (6) | 2 (2) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 2 (2) | 5 (5)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 4 (5) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 5 (5) | 6 (6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (6) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 4 (5) | 4 (4) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 3 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The steering committee will be responsible for the publication and presentation strategy. All publications will be based on data released or agreed by Bayer, verified by the steering committee.